CLINICAL TRIAL: NCT03228329
Title: Validation of Electrical Cardiometry in Resuscitation of Patients Undergoing Orthotopic Liver Transplantation
Brief Title: Validation of Cardiometry in Resuscitation of Patients Undergoing Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Elayashy Mohamed Ahmed Hassan, clinical professor, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: N-43-2017
Record Dates: First submitted 2017-07-13; First posted 2017-07-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Liver Transplantation
Keywords: cardiometry; stroke volume; liver transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cardiometry (Other): fluid boluses will be given when there will be hypovolemia assessed by presence of pulse pressure variations
  Interventions: Other: fluid boluses

INTERVENTIONS:
Other: fluid boluses — fluid boluses will be given when there will be hypovolemia assessed by presence of pulse pressure variations

SUMMARY:
aim of our study to validate electrical cardiometry readings against same readings by transoesophageal echo. we will validate stroke volume (SV) readings stroke volume variation(SVV), index of contractility.

DETAILED DESCRIPTION:
Induction of anaesthesia will be by using propofol (2mg.kg) IV, fentanyl (1-2μg. kg) IV and atracurium (0.5 mg.kg) IV. Anaesthesia will be maintained with Sevoflurane adjusted between 1-2% in an air ⁄ oxygen mix (FiO2 0.6), fentanyl infusion at 1-2 μg.kg/h and atracurium infusion at 0.5 mg.kg/ h. Mechanical ventilation will be provided by using a Dräger anaesthesia machine (Dräger Primus®, Germany) using a tidal volume of 6-8 ml.kg with the respiratory rate adjusted to maintain the PaCO2 between 4-4.6 kilopascal (kPa) and positive end expiratory pressure (PEEP) of 5 cmH2O. All patients will be monitored for five lead ECG, peripheral oxygen saturation, noninvasive and invasive arterial blood pressure, temperature, end-tidal carbon dioxide tension, hourly urinary output, and central venous pressure (CVP). A 7-Fr triple lumen CVP catheter (Arrow International Inc, Reading, PA, USA) will be inserted into the right internal jugular vein.

All patients will receive 6ml /kg/h Ringer acetate solution as a maintenance intraoperative fluid. If SVV is more than 15%, the patient will be considered as fluid responder and will receive a 250-ml bolus of albumin 5% to maintain SVV ≤15%. Blood transfusion will be given based on a hemoglobin level (< 7 g/dl). Norepinephrine will be administered if the mean arterial pressure was less than 70 mmHg. Epinephrine will be administered if mean arterial blood pressure was less than 70 mm Hg and the cardiac index was less than 2.5 L/min/m2 despite sufficient volume infusion, to maintain a target cardiac index of 2.5-3.0 L/min/m2

Electrical cardiometry (EC) Examination:

1. ECG electrodes will be placed on the bare skin of patients in the following positions:

   1. On the left neck below the ear;
   2. Directly above the midpoint of the left clavicle;
   3. Along the left mid-axillary line at the level of the xiphoid process;
   4. Two inches caudal from the third electrode.
2. Patient characteristics of sex, age, height and weight will be entered into the monitor.
3. Clocks on the EC and trans esophageal echo (TEE) machine will be synchronized prior to data collection.
4. The EC monitor will be programmed to capture moving averages of variables based on the previous 10 cardiac cycles and to record those averages every10 s.
5. Only EC data with a signal quality index (SQI) of >70 will be included in the analysis.

Echo Examination:

1. A single LVOT diameter will be measured for each patient as the distance between the inﬂection points at the base of the aortic valve cusps from the left ventricle long axis view during systole.
2. Assuming a circular cross section, the LVOT area will be calculated from the LVOT diameter as:

   π X (LVOT diameter/ 2)2 = (LVOT diameter)2 X 0.785
3. Pulse wave Doppler sampling cursor will be placed in the middle of the LVOT immediately proximal to the aortic valve in 5 chamber deep transgastric view.
4. The sonographer manually will trace the velocity-time envelope.
5. SV values will be identified for 10 cycles and averaged to obtain SV-Doppler max and SV-Doppler min. The mean SV (SV-Doppler mean) will be calculated as (SV-Doppler max - SV-Doppler min)/2.
6. SVV-Doppler will be calculated as (SV-Doppler max - SV-Doppler min)/SV-Doppler mean.
7. Peak aortic velocity, time to peak and mean acceleration will be calculated.

Mini Fluid challenge:

1. Mini fluid challenge will be done by 150 cc crystalloid over 1 min
2. 2 sets of measurement of SV and SVV will be obtained

   1. The first set of measurement will be obtained before fluid challenge.
   2. The second set will be obtained immediately after fluid challenge. Other data will be recorded as;heart rate (HR), systolic BP, Diastolic BP, mean BP, CVP and pulse pressure variation (PPV)

ELIGIBILITY:
Inclusion Criteria:

* ASA II to IV patients with end-stage liver disease
* patients undergoing orthotopic living donor liver transplantation
* age > 18 years

Exclusion Criteria:

* acute fulminant liver failure
* age < 18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
stroke volume | 5 minutes after reperfusion.
  record stroke volume assessed by noninvasive cardiometry and TEE
stroke volume | 15 minutes after dissection phase.
  record stroke volume assessed by noninvasive cardiometry and TEE

SECONDARY OUTCOMES:
stroke volume variation | 5 minutes after reperfusion.
  record stroke volume assessed by noninvasive cardiometry and TEE
stroke volume variation | 15 minutes after dissection phase
  record stroke volume variation assessed by noninvasive cardiometry and TEE

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mohamed mokhtar, M.D, Study Director — kasralainy faculty of medicine, Cairo university
Locations (1):
- Kasr Alainy Hospital , Faculty of Medicine, Cairo, Egypt

REFERENCES:
- [Background] Bechstein WO, Neuhaus P. [Bleeding problems in liver surgery and liver transplantation]. Chirurg. 2000 Apr;71(4):363-8. doi: 10.1007/s001040051066. German. PMID 10840602
- [Background] Rossi G, Langer M, Maggi U, Reggiani P, Caccamo L, Gatti S, Paone G, Vannelli A, Prato P, Doglia M, Melada E, Latham L, Fassati LR. Veno-venous bypass versus no bypass in orthotopic liver transplantation: hemodynamic, metabolic, and renal data. Transplant Proc. 1998 Aug;30(5):1871-3. doi: 10.1016/s0041-1345(98)00465-5. No abstract available. PMID 9723316
- [Background] Bulkley GB. Reactive oxygen metabolites and reperfusion injury: aberrant triggering of reticuloendothelial function. Lancet. 1994 Oct 1;344(8927):934-6. doi: 10.1016/s0140-6736(94)92276-4. No abstract available. PMID 7848422
- [Derived] Mukhtar AM, Elayashy M, Sayed AH, Obaya GM, Eladawy AA, Ali MA, Dahab HM, Khalaf DZ, Mohamed MA, Elfouly AH, Behairy GM, Abdelaal AA. Validation of electrical velocimetry in resuscitation of patients undergoing liver transplantation. Observational study. J Clin Monit Comput. 2020 Apr;34(2):271-276. doi: 10.1007/s10877-019-00313-z. Epub 2019 Apr 19. PMID 31004273